CLINICAL TRIAL: NCT02506244
Title: mHealth Screening to Prevent Strokes (mSToPS)
Brief Title: mHealth Screening to Prevent Strokes
Acronym: mSToPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); Aetna, Inc. (Industry)
Responsible Party: Principal Investigator, Steven Steinhubl, Director, Digital Medicine, Scripps Translational Science Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Version 3.5
Record Dates: First submitted 2015-07-17; First posted 2015-07-23 (Estimated); Results first posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Wearable device; Wristband; ECG Patch; Strokes; Asymptomatic; Heart Rhythm; Home Monitoring
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Immediate Monitoring (Experimental): Individuals randomized to immediate monitoring will receive the ZIO XT patch sensor and wear it for the first and last 2 week period of the 4 month monitoring period of time 0 to 4 months.
  Note: Approximately 250 consenting participants will also be invited to participate in a sub-study to wear an additional monitoring device (Amiigo wristband) continuously over the 4 month monitoring period.
  Interventions: Device: iRhythm ZIO XT Patch; Device: Wristband by Amiigo
- Delayed Monitoring (Active Comparator): Individuals randomized to delayed monitoring will receive usual care for 4 months after which they will receive the ZIO XT patch sensor and wear it for the first and last 2 week period of study months 4 through 8.
  Note: Approximately 250 consenting participants will also be invited to participate in a sub-study to wear an additional monitoring device (Amiigo wristband) daily for months 4 through 8.
  Interventions: Device: iRhythm ZIO XT Patch; Device: Wristband by Amiigo

INTERVENTIONS:
Device: iRhythm ZIO XT Patch — Single-lead ECG monitoring via a wearable patch
Device: Wristband by Amiigo — Determines pulse rate using photoplethysmography.

SUMMARY:
The purpose of this study is to investigate whether it is possible to identify a high-risk cohort suitable for screening for asymptomatic atrial fibrillation using claims data, and then engage those individuals in a mobile health technology-enabled home monitoring program in order to document previously undiagnosed atrial fibrillation, and provide clinical evidence of an outcomes benefit associated with this early detection.

DETAILED DESCRIPTION:
The purpose of this study is to propose to study two different methods of intermittent rhythm monitoring in a cohort of individuals without prior history of atrial fibrillation, but determined to be at increased risk based on clinical risk factors, and compare the rate of atrial fibrillation detection through monitoring relative to routine care.

ELIGIBILITY:
Participants:

The study population will be derived from the Aetna and Medicare populations.

Inclusion Criteria:

* Male or females age > 75 or
* Male age > 55, or females age > 65, and
* Prior CVA, or
* Heart failure, or
* Diagnosis of both diabetes and hypertension, or
* Mitral valve disease, or
* Left ventricular hypertrophy, or
* COPD requiring home O2, or
* Sleep apnea, or
* History of pulmonary embolism, or
* History of myocardial infarction, or
* Diagnosis of obesity

Exclusion Criteria:

* Current or prior diagnosis of atrial fibrillation, atrial flutter or atrial tachycardia
* Receiving chronic anticoagulation therapy
* Hospice care
* End stage renal disease
* Diagnosis of moderate or greater dementia
* Implantable pacemaker and/or defibrillator
* History of skin allergies to adhesive patches
* Known metastatic cancer
* Aetna Compassionate Care Program (ACCP) participants - individuals with advanced illness and limited life expectancy

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6135 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Steinhubl, Principal Investigator — Study Principal Investigator
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reynolds MR, Stein AB, Sun X, Hytopoulos E, Steinhubl SR, Cohen DJ. Cost-Effectiveness of AF Screening With 2-Week Patch Monitors: The mSToPS Study. Circ Cardiovasc Qual Outcomes. 2023 Nov;16(11):e009751. doi: 10.1161/CIRCOUTCOMES.122.009751. Epub 2023 Oct 31. PMID 37905421
- [Derived] Steinhubl SR, Waalen J, Sanyal A, Edwards AM, Ariniello LM, Ebner GS, Baca-Motes K, Zambon RA, Sarich T, Topol EJ. Three year clinical outcomes in a nationwide, observational, siteless clinical trial of atrial fibrillation screening-mHealth Screening to Prevent Strokes (mSToPS). PLoS One. 2021 Oct 5;16(10):e0258276. doi: 10.1371/journal.pone.0258276. eCollection 2021. PMID 34610049
- [Derived] Baca-Motes K, Edwards AM, Waalen J, Edmonds S, Mehta RR, Ariniello L, Ebner GS, Talantov D, Fastenau JM, Carter CT, Sarich TC, Felicione E, Topol EJ, Steinhubl SR. Digital recruitment and enrollment in a remote nationwide trial of screening for undiagnosed atrial fibrillation: Lessons from the randomized, controlled mSToPS trial. Contemp Clin Trials Commun. 2019 Jan 7;14:100318. doi: 10.1016/j.conctc.2019.100318. eCollection 2019 Jun. PMID 30656241
- [Derived] Steinhubl SR, Waalen J, Edwards AM, Ariniello LM, Mehta RR, Ebner GS, Carter C, Baca-Motes K, Felicione E, Sarich T, Topol EJ. Effect of a Home-Based Wearable Continuous ECG Monitoring Patch on Detection of Undiagnosed Atrial Fibrillation: The mSToPS Randomized Clinical Trial. JAMA. 2018 Jul 10;320(2):146-155. doi: 10.1001/jama.2018.8102. PMID 29998336

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an observational study with two study arms, an immediate monitoring group and a delayed monitoring group. This was not a cross-over design study. The control group for this study consisted of participants that were not given the Zio patch. This group was used to compare who got routine care compared to the other arms that received the Zio patches.
Groups:
- Immediate Monitoring: Individuals randomized to immediate monitoring will receive the ZIO XT patch sensor and wear it for the first and last 2 week period of the 4 month monitoring period of time 0 to 4 months.
  Note: Approximately 250 consenting participants will also be invited to participate in a sub-study to wear an additional monitoring device (Amiigo wristband) continuously over the 4 month monitoring period.
  iRhythm ZIO XT Patch: Single-lead ECG monitoring via a wearable patch
  Wristband by Amiigo: Determines pulse rate using photoplethysmography.
- Delayed Monitoring: Individuals randomized to delayed monitoring will receive usual care for 4 months after which they will receive the ZIO XT patch sensor and wear it for the first and last 2 week period of study months 4 through 8.
  Note: Approximately 250 consenting participants will also be invited to participate in a sub-study to wear an additional monitoring device (Amiigo wristband) daily for months 4 through 8.
  iRhythm ZIO XT Patch: Single-lead ECG monitoring via a wearable patch
  Wristband by Amiigo: Determines pulse rate using photoplethysmography.
- Match Controls: Observational matched controls that underwent routine care and were not given a Zio patch
Period: Overall Study
Arm/Group | Immediate Monitoring | Delayed Monitoring | Match Controls
Started | 1366 | 1293 | 3476
Completed | 908 | 834 | 3476
Not Completed | 458 | 459 | 0
Not completed — Did not undergo active monitoring | 458 | 459 | 0

BASELINE CHARACTERISTICS:
Groups:
- Matched Controls: Individuals that underwent routine care and were not given a Zio XT patch sensor.
- Total: Total of all reporting groups
Arm/Group | Immediate Monitoring | Delayed Monitoring | Matched Controls | Total
Number analyzed (Participants) | 1366 | 1293 | 3476 | 6135
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (7.4) | 73.1 (7.2) | 73.7 (7.0) | 73.7 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 521 | 505 | 1408 | 2434
  Male | 845 | 788 | 2068 | 3701
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1366 | 1293 | 3476 | 6135

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Newly Diagnosed AF in the Immediate vs Delayed Monitoring Group
Description: Incidence of newly diagnosed AF as defined by at least 30 seconds of AF or atrial flutter at the end of the 4 month monitoring period compared to the delayed monitoring cohort (primary) and observational control (secondary)
Time Frame: End of 4 month monitoring period
Population: In the intention-to-treat analysis of the randomized clinical trial, we analyzed the incidence of new AF cases in the immediate monitoring group vs the delayed monitoring groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Monitoring | Delayed Monitoring
Number analyzed (Participants) | 1366 | 1293
Participants | 53 | 12

2. Secondary Outcome: Prevalence of Atrial Fibrillation in Both Monitoring Groups Versus the Matched Controls
Description: In the observational study, over 12 months of follow-up, we looked at the prevalence of AF in the actively monitored and delayed monitored cohorts.
Time Frame: 1 year
Population: 906 participants that were in the immediate monitoring group had 12 months of follow-up data, 832 participants in the delayed monitoring group had 12 months of follow-up data
Measure: Count of Participants; unit: Participants
Groups:
- Immediate Monitoring: Individuals randomized to immediate monitoring will receive patch in first 4 months
- Matched Controls: Observational control cohort that was not given a Zio patch, but instead underwent routine care
Arm/Group | Immediate Monitoring | Delayed Monitoring | Matched Controls
Number analyzed (Participants) | 906 | 832 | 3476
Participants | 63 | 46 | 81

ADVERSE EVENTS:
Time Frame: 1 year
Description: The only adverse events reported in this study were in relation to skin irritations developed from wearing the Zio patch. There was no risk of all-cause mortality or serious adverse events connected to wearing the patch so all-cause mortality and serious adverse events were not monitored/assessed The observational controls did not receive a patch and thus were not actively monitored for adverse events.
Arm/Group | Immediate Monitoring | Delayed Monitoring
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 20/908 | 21/834
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Immediate Monitoring (N=908) | Delayed Monitoring (N=834)
Skin irritation from Zio XT patch (Skin and subcutaneous tissue disorders) | 20 (20) | 21 (21) — Minor skin irritation that resulted from wearing the patch. All resolved.
Skin irritation from Amigo wristband (Skin and subcutaneous tissue disorders) | 0/230 (0) | 0/230 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT02506244/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/44/NCT02506244/SAP_001.pdf